CLINICAL TRIAL: NCT04223076
Title: Clinical Performance of Two 0.2% Chlorhexidine Mouth Rinses After Periodontal Surgery. A Blinded, Intra-individual Cross-over Clinical Trial
Brief Title: Clinical Effect of Chlorhexidine Mouthwash After Periodontal Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Erik Mauland, DDS, University of Oslo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2020/121314
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Periodontal Diseases; Periodontitis; Dental Plaque
Keywords: Periodontal Index
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Dental Plaque | interventions — Chlorhexidine

STUDY DESIGN:
Intervention Model Description: Intra individual cross-over, double intervention
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chlorhexidine 0.2% mouthwash control (Experimental): Chlorhexidine 0.2%, Corsodyl Intervention rinsing 60 sec twice daily
  Interventions: Drug: Chlorhexidine 0.2%, Corsodyl
- Chlorhexidine 0.2% mouthwash with an Anti Discoloring System (Experimental): Chlorhexidine 0.2%, Curasept Intervention rinsing 60 sec twice daily
  Interventions: Drug: Chlorhexidine 0.2%, Curasept

INTERVENTIONS:
Drug: Chlorhexidine 0.2%, Corsodyl — Comparison of Corsodyl and Curasept
  Arms: Chlorhexidine 0.2% mouthwash control
Drug: Chlorhexidine 0.2%, Curasept — Chlorhexidine 0.2% mouthwash with an Anti Discoloring System (ADS)
  Arms: Chlorhexidine 0.2% mouthwash with an Anti Discoloring System

SUMMARY:
Chlorhexidine is the gold standard of dental plaque prevention. Recent research have demonstrated that 0.2% Chlorhexidine solutions are more effective than 0.12% and 0.06% Chlorhexidine solutions. Several 0.2% solutions are available on the market. This study aimed to compare effectiveness of two commercially available 0.2% chlorhexidine mouthwashes. Patients, that after initial periodontal therapy, had a need for two periodontal surgeries, will be invited to join. After one surgical session, the patient will receive one 0.2% chlorhexidine solution, and after the next surgical session the patient will receive the other 0.2% chlorhexidine solution. Plaque and gingivitis will be recorded, as well as side effects.

ELIGIBILITY:
Inclusion Criteria:

Periodontitis, stage III and IV

Exclusion Criteria:

Uncontrolled diabetes Systemic conditions associated with excessive bleeding Uncontrolled hypertension

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Plaque index | 14 days intervention period
  Dental Plaque
Gingival Index | 14 days intervention period
  Gingivitis

CONTACTS AND LOCATIONS:
Overall Officials: Anne Merete Aass, Professor, Study Chair — University of Oslo
Locations (1):
- Erik Mauland, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes